CLINICAL TRIAL: NCT05484960
Title: Multicenter Collection of Uniform Data on Patients With Cognitive Impairment in the Philippines: the Philippine Neurological Association One Database -Dementia (PNA1DB-Dementia)
Brief Title: The Philippine Neurological Association One Database -Dementia
Acronym: PNA1DB-Dem
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philippine Neurological Association (Other)
Collaborators: University of Santo Tomas Hospital, Philippines (Other); Baguio General Hospital and Medical Center, Philippines (Unknown); East Avenue Medical Center, Philippines (Other Government); Jose R. Reyes Memorial Medical Center (Other Government); Makati Medical Center (Other); Quirino Memorial Medical Center, Philippines (Unknown); St. Luke's Medical Center, Philippines (Other); The Medical City, Philippines (Other); University of the East- Ramon Magsaysay Memorial Medical Center, Philippines (Unknown); University of the Philippines Manila - Philippine General Hospital (Other); Chong Hua Hospital, Philippines (Unknown)
Responsible Party: Sponsor
Other Study IDs: PNA2020_0X
Record Dates: First submitted 2022-07-17; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Impairment; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cognitive assessment — The clinical diagnosis will be made based on the criteria set by the investigators. Clinical history and bedside objective assessment in the form of Montreal Cognitive Assessment-Philippines (MoCA-P) or Mini Mental Status Examination-Philippines (MMSE-P), supported by a neuroimaging study (if neuroimaging is not done, diagnosis will be supported by the Hachinski Ischemic Score).

SUMMARY:
This is a pragmatic, multi-center, prospective, observational, non-interventional study and standing database of patients seen at the training institution for cognitive impairment diagnosed with Mild Cognitive Impairment (MCI) or Dementia.

All patients seen at the training institution clinically diagnosed with MCI or dementia by their neurologists will be invited to participate in the study. The investigators will confirm the diagnosis and will explain the study as well as the patient information sheet to the patient and/or legal representative. All eligible patients seen will be assigned a study identification number. Data will be collected by the investigators as the patient undergoes routine clinical evaluation. Corresponding anonymized data on demographics, medical history and risk factors, level of functional impairment, diagnosis, baseline cognitive scores and management will be collected from each patient and entered in the database using a secure online data collection tool.

DETAILED DESCRIPTION:
The investigators will confirm the diagnosis and will explain the study as well as the patient information sheet to the patient and/or legal representative. All eligible patients seen will be assigned a study identification number. Data will be collected by the investigators as the patient undergoes routine clinical evaluation. Corresponding anonymized data on demographics, medical history and risk factors, level of functional impairment, diagnosis, baseline cognitive scores and management will be collected from each patient and entered in the database using a secure online data collection tool. Patients who withdraw participation verbally or in writing are excluded by the investigator from further participation. Withdrawal from the study will be properly documented, including date, time, and reason for withdrawal. Withdrawn subjects will not have their clinical data included in the database.

Collective data will be extracted, summarized, and analyzed every year with oversight provided by the Philippine Neurological Association (PNA). To be able to assess trends and changes over time, data collection for this study will span 3 years from study initiation, after which the utility of an extension or a re-implementation of the study will be assessed by the PNA.

ELIGIBILITY:
Inclusion Criteria

* Patient with cognitive impairment diagnosed with Mild Cognitive Impairment or Dementia.
* 18 years old or older.
* Must be a Filipino Citizen.
* Seen and evaluated in the participating hospital by a neurologist.
* If required by the institutional review board/ethics committee, signed or verbal informed consent for participation in the study from the patient or a legal representative.

Exclusion Criteria

• Any condition which, in the study investigator's opinion, may jeopardize the patient by his/her participation in this study or affect the validity of the study results.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen and evaluated at the participating sites are eligible to be included in the study if they fulfill all inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of dementia and mild cognitive impairment in the study population | on Day 1
  To determine the frequency of dementia and mild cognitive impairment in the study

SECONDARY OUTCOMES:
F frequency of the different types of dementia in the study population | on Day 1
  To determine the frequency of the different types of dementia in the study population using the clinical diagnosis
Frequency of risk factors for dementia in the study population | on Day 1
  o determine the frequency of risk factors for dementia in the study population. (age, sex, educational attainment, family history, physical activity, smoking history, alcohol consumption, cardiovascular and cerebrovascular risk factors, chemical exposure, substance abuse, previous psychiatric condition and hearing impairment)
Demographic characteristics of patients with dementia or mild cognitive impairment | on Day 1
  To describe the demographic characteristics of patients with dementia or mild cognitive impairment as to age at the time of diagnosis, age of onset of symptoms, sex, level of income (of patient or caregiver), location of clinic or hospital, current or previous occupation, educational attainment, neurologic exam findings
Dementia Severity | on Day 1
  To categorize dementia severity in each subtype as mild, moderate and severe based on the initial MMSE score at the time of diagnosis.
Diagnostic tests used at the time of the diagnosis | on Day 1
  To describe the types of diagnostic tests commonly done at the time of diagnosis, such as neuroimaging, blood tests, EEG
Pharmacologic and nonpharmacologic modalities used | on Day 1
  To identify pharmacologic and nonpharmacologic modalities of treatment currently being used in the treatment of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Ma. Lourdes C Joson, MD, Principal Investigator — Philippine Neurological Association
Locations (11):
- Philippines (11):
  - Baguio General Hospital and Medical Center, Baguio City, Baguio
  - Chong Hua Hospital, Cebu City, Cebu
  - Makati Medical Center, Makati City, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - East Avenue Medical Center, Quezon City, National Capital Region
  - Quirino Memorial Medical Center, Quezon City, National Capital Region
  - St. Luke's Medical Center, Quezon City, National Capital Region
  - Jose R. Reyes Memorial Medical Center, Manila
  - University of Santo Tomas Hospiatl, Manila
  - University of the East- Ramon Magsaysay Memorial Medical Center, Manila
  - University of the Philippines - Philippine General Hospital, Manila

IPD SHARING:
Plan to Share IPD: No
To be available upon request